CLINICAL TRIAL: NCT04776031
Title: Evaluation of the R:GEN Laser System as an Intervention in Subjects With Early Stages of Age Related Macular Degeneration (AMD) for Safety and Exploratory Efficacy Outcomes
Brief Title: Evaluation of R:GEN as Intervention in Subjects With Early Stages of AMD for Safety and Exploratory Efficacy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lutronic Vision, Inc (Industry)
Collaborators: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56173
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Early Age Related Macular Degeneration (Disorder)
Keywords: Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; High risk early age related macular degeneration; Laser Treatment
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laser Treatment (Experimental): Laser treatment using the R:GEN Laser System on Day 1 and at Week 24
  Interventions: Device: R:GEN Laser System

INTERVENTIONS:
Device: R:GEN Laser System — Laser Treatment

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the R:GEN Laser System in subjects with the early stages of age-related macular degeneration.

DETAILED DESCRIPTION:
This clinical study is a prospective, single-center, single-arm, open-label, pilot study to evaluate the safety and tolerability of the R:GEN Laser System and to collect information on the severity of AMD in subjects with bilateral large drusen. All participants will receive the intervention at the baseline visit and at the 24-week visit. All participants will be evaluated at 24 and 48 weeks from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years and over
* Best Corrected Visual Acuity [BCVA] of 6/12 [20/40] or better in each eye
* Bilateral large drusen: at least 1 druse ≥125 µm in each eye within an inner macular zone [a circle with a radius of 1500 µm centered on the fovea], and with or without pigment;
* Ability and willingness to consent, receive laser treatment, and complete all visits

Exclusion Criteria:

* Any evidence of definite reticular pseudo drusen [RPD] > 2-disc areas [DAs] as seen either by fundus autofluorescence [FAF] or near-infrared reflectance [NIR] enface imaging in each eye
* Any evidence of geographic atrophy [GA] within the macula [a circle with a radius of 3000 microns centered on the fovea] excluding peripapillary atrophy
* Any evidence of nascent GA, or worse evidence of atrophy (complete RPE and outer retinal atrophy) as determined by OCT: including the subsidence of the inner nuclear layer and outer plexiform layer [OPL], or the presence of a hyporeﬂective wedge-shaped band within the limits of the OPL, and accompanied by attenuation or absence of the RPE and hypertransmission into the choroid
* Current choroidal neovascularization [CNV], (determined on multimodal imaging [MMI], but angiogram not required) or past evidence of CNV, including the presence of non-exudative macular neovascularization [NE-MNV] [determined by OCT-A]
* Asymptomatic sub-retinal fluid [SRF] [a slither < 50 µm allowed]
* Any current ocular disease or condition in the study eye including diseases affecting the optic nerve, the anterior chamber, and autoimmune or systemic inflammatory conditions in which there are ocular manifestations that either are undergoing or require treatment, or history of ocular disease within 3 months of screening
* A central macular serous pigment epithelial detachment greater than 1000 µm in diameter; a central macular drusenoid detachment > 1000 µm with hyper reflective foci [HRF] and hypertransmission; or any central macular drusenoid pigment epithelial detachments >2000 µm
* Previous retinal or ocular surgery within 3 months prior to screening, the effects of which may now or in the future complicate assessment of AMD
* Any history of prior laser treatment to the retina
* Any systemic medication known to be toxic to the retina
* Known hypersensitivity to fluorescein or indocyanine green
* Sensitivity to application of a contact lens
* History or presence of uncontrolled glaucoma, ocular hypertension, or intraocular pressure > 24 mmHg
* Cataract which in the opinion of the investigator limits evaluation of the retina or requires cataract surgery within 12 months
* Pregnant or lactating women
* Subject who is currently in a clinical study, or has received other active investigational therapy, within 30 days of the screening visit
* Subject who is considered ineligible for this study in the investigator's medical judgment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
To access the safety and tolerability of the R:GEN Laser System in subjects with the early stages of AMD. | up to 48 weeks
  Incidences of Serious Adverse Events, Serious Adverse Device Effects, Unanticipated Serious Adverse Device Effects

SECONDARY OUTCOMES:
To evaluate the progression in severity of AMD after treatment with the R:GEN Laser System at 24 weeks and 48 weeks post-treatment. | 24 weeks and 48 weeks post-treatment
  Evidence of the presence of late AMD

CONTACTS AND LOCATIONS:
Overall Officials: Robyn H Guymer, MBBS, PhD, Principal Investigator — Center for Eye Research Australia
Locations (1):
- Centre for Eye Research Australia - Royal Victorian Eye & Ear Hospital, East Melbourne, Victoria, Australia